CLINICAL TRIAL: NCT04485702
Title: A Pilot Phase 1, Randomized, Single-Dose, 6-Sequences, 3-Period, Crossover Bioavailability Study of MELT-100 (Midazolam and Ketamine Sublingual Tablet) and Intravenous Midazolam or Ketamine in Healthy Volunteers
Brief Title: Phase 1 Bioavailability Study of MELT-100 (Midazolam and Ketamine Sublingual) and IV Midazolam or Ketamine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Melt Pharmaceuticals (Industry)
Collaborators: Worldwide Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: MELT-100-001
Record Dates: First submitted 2020-07-17; First posted 2020-07-24 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Intervention Model Description: Randomized, Single-Dose, 6-Sequence, 3-Period, Crossover
Who Masked: Participant
Masking Description: randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- MELT-100 (Active Comparator): 3mg midazolam and 25mg ketamine sublingual tablet
  Interventions: Drug: MELT-100
- IV midazolam (Active Comparator): 2mg Intravenous midazolam
  Interventions: Drug: Midazolam injection
- IV ketamine (Active Comparator): 6mg Intravenous ketamine
  Interventions: Drug: Ketamine Injectable Product

INTERVENTIONS:
Drug: Midazolam injection — 2mg IV
  Arms: IV midazolam
Drug: Ketamine Injectable Product — 6mg IV
  Arms: IV ketamine
Drug: MELT-100 — midazolam 3mg and ketamine 25mg SL tablet
  Arms: MELT-100

SUMMARY:
Comparative Bioavailability study testing MELT-100 (midazolam and ketamine sublingual tablet) and IV midazolam or ketamine in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* A subject must satisfy all of the following criteria to be eligible for study participation:

  1. Able to understand and voluntarily consent to participation in this study, and provides written informed consent before the start of any study-specific procedures.
  2. Healthy adult male or female ≥55 years of age.
  3. Normally active and otherwise judged to be in good health on the basis of medical history and physical examination.
  4. Has vital signs (measured sitting after a minimum 3 minutes rest) at Screening within the following ranges: heart rate: 40-100 bpm; systolic blood pressure (BP): 90-145 mmHg; diastolic BP: 50-95 mmHg. Out-of-range vital signs may be repeated once.
  5. Has a body temperature ≤37.7 degrees C
  6. Body weight ≥55 kg
  7. Body mass index (BMI) 18.0 to 32.0 kg/m2 (inclusive)
  8. Female subjects are eligible only if the following applies:

     Surgically sterile (bilateral tubal ligation, hysterectomy, or bilateral oophorectomy), or postmenopausal (confirmed with serum FSH at Screening)
  9. Male subjects must either be surgically sterile (vasectomy at least 3 months prior to first dose) or agree to use an acceptable method of birth control (see Section 4.4) from Screening through EOS.
  10. Is willing and able to remain in the study unit for the entire duration of each confinement period.

Exclusion Criteria:

* Subjects will be excluded from study participation for any of the following:

  1. History or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, ophthalmologic, dermatologic, neurologic, oncologic, or psychiatric disease or any other condition that, in the opinion of the Investigator, would jeopardize the safety of the subject or the validity of the study results.
  2. Has a history of glaucoma, asthma, chronic obstructive pulmonary disease, or thyroid disease.
  3. Clinically significant illnesses within 4 weeks of the administration of study medication (including flu, flu-like symptoms, diarrhea, vomiting, fever, sore throat) or acute illness at the time of either the pre-study medical evaluation or dosing.
  4. Has been in contact with someone within the last month who has tested positive for SARS-CoV-2.
  5. Clinically significant surgery within 4 weeks prior to the administration of the study medication.
  6. Has participated in another clinical trial (randomized subjects only) within 30 days before the first dose of study medication.
  7. An active malignancy of any type, or has been diagnosed with cancer within 5 years prior to Screening (excluding squamous or basal cell carcinoma of the skin).
  8. History or presence of allergic or adverse response to midazolam, ketamine, Versed, KETALAR, or any ingredients of MELT-100 or related drugs.
  9. Use of any over-the-counter (OTC) medication (including nutritional or dietary supplements, herbal preparations, or vitamins) within 7 days before the first dose of study medication until the EOS without evaluation and approval by the Investigator.
  10. Use of any prescription medication, except statin drugs or hormonal replacement therapy, from 14 days before the first dose of study medication until the EOS without evaluation and approval by the Investigator.
  11. Have had a depot injection or an implant of any drugs 3 months prior to administration of study medication.
  12. Has been treated with any known drugs that are moderate or strong inhibitors/inducers of cytochrome P450 (CYP) enzymes (e.g., barbiturates, phenothiazines, cimetidine, carbamazepine) within 30 days before the first dose of study medication, and that, in the Investigator's judgment, may impact subject safety or the validity of the study results.

      Specifically, the use of any drugs known to inhibit CYP2C9 and CYP3A4 enzymes (examples include amiodarone, fluconazole, ketoconazole, itraconazole, clarithromycin, ritonavir, erythromycin, grapefruit or orange or apple juice) or any drugs that are highly protein-bound (for example, warfarin, cyclosporine, amphotericin B) within 30 days prior to the first dose of study medication, and that in the Investigator's judgment may impact subject safety or the validity of the study results.
  13. Blood or plasma donation within 30 days before the first dose of study medication until the EOS. It is recommended that blood/plasma donations not be made for at least 30 days after the EOS.
  14. Has any prior history of substance abuse or treatment (including alcohol).

      1. History of significant alcohol abuse within 6 months of Screening or any indication of the regular use of more than 2 units of alcohol per day (1 unit = 50 mL of wine or 360 mL of beer or 45 mL of alcohol 40%).
      2. History of use of marijuana within 3 months of Screening or drugs such as cocaine, phencyclidine (PCP), within 1 year of Screening.
  15. Smoking or use of tobacco- or nicotine-containing products within 60 days before the first dose of study medication until the EOS Note: Nonsmokers are preferred for this study.
  16. Any food allergy, intolerance, restriction, or special diet that, in the opinion of the Investigator, contraindicates the subject's participation in this study.
  17. Has been on a significantly abnormal diet during the 4 weeks preceding the first dose of study medication.
  18. Consumption of beverages or foods that contain alcohol, grapefruit, poppy seeds, broccoli, Brussels sprouts, pomegranate, star fruit, char-grilled meat, or caffeine/xanthine from 48 hours before the first dose of study medication until the EOS. Subjects will be instructed not to consume any of the above products; however, allowance for an isolated single incidental consumption may be evaluated and approved by the study Investigator based on the potential for interaction with the study drug.
  19. Engagement in strenuous exercise from 48 hours before the first dose of study medication until the EOS.
  20. A clinically significant abnormal finding on the physical examination, medical history, electrocardiogram (ECG), or clinical laboratory results at Screening.

      Note: Laboratory test values above or below the normal range does not necessarily indicate that the value is "clinically significant." The determination should be made at the discretion of the Investigator with consultation, when necessary, with the Sponsor.
  21. Presence of active infection, mucositis, cold sores, apthous ulcers, vesicles, viral lesions, local irritation/inflammation, or periodontal disease of the oral cavity. In addition, evidence of piercings of the tongue or anywhere in the oral cavity, history of oral cavity piercings, or history of significant dental disease or braces or oral hardware.
  22. Clinically significant ECG abnormalities at Screening.
  23. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels ˃1.25 times the upper limit of normal at Screening or Check-in for Period 1.
  24. Is a female with a positive pregnancy test result.
  25. Has a positive urine screen for drugs of abuse (amphetamines, barbiturates, benzodiazepines, cocaine, cannabinoids, opiates) or cotinine.
  26. Has a positive test for hepatitis B surface antigen, hepatitis C antibody, or human immunodeficiency virus (HIV) at Screening or has been previously treated for hepatitis B, hepatitis C, or HIV infection.
  27. Has poor venous access during blood sampling at Screening.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2020-08-29 (Actual); Study Completion 2020-08-29 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 24 hours
Area under the plasma concentration versus time curve (AUC) | 24 hours
Time to peak plasma concentration (Tmax) | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Zamora, MD, Principal Investigator — Worldwide Clinical Trials
Locations (1):
- WWCT, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No